CLINICAL TRIAL: NCT04534218
Title: Regorafenib in Combination With Metronomic Cyclophosphamide, Capecitabine, and Low-dose Aspirin in Metastatic Colorectal Cancer Carcinoma An Open-label Phase II
Brief Title: Regorafenib in Combination With Metronomic Chemotherapies, and Low-dose Aspirin in Metastatic Colorectal Cancer
Acronym: REPROGRAM-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/490
Record Dates: First submitted 2020-07-16; First posted 2020-09-01 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Colo-rectal Cancer; Metastatic Cancer
Keywords: regorafenib; metronomic chemotherapy; colon cancer
MeSH Terms: conditions — Colonic Neoplasms; Neoplasm Metastasis | interventions — regorafenib; Cyclophosphamide; Capecitabine; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): REGORAFENIB:
  * For the first cycle: regorafenib will be administered according to the "REDOS" schedule (80 mg daily for week 1, 120 mg daily for week 2 and 160 mg daily for the third week of the first cycle).
  * For the following cycles: regorafenib will be administered at a 80, 120 or 160 mg daily dose according to toxicity observed with the last dose used in the first cycle.
  METRONOMIC CHEMOTHERAPIES:
  * Capecitabine: 625mg/m²/orally twice daily continuously for 6 months
  * Cyclophosphamide: 50 mg per os, daily, for 6 months
  ASPIRIN:
  75 mg orally and daily until progression
  Interventions: Drug: Regorafenib; Drug: Cyclophosphamide; Drug: Capecitabine; Drug: Aspirin

INTERVENTIONS:
Drug: Regorafenib — * For the first cycle: regorafenib will be administered according to the "REDOS" schedule (80 mg daily for week 1, 120 mg daily for week 2 and 160 mg daily for the third week of the first cycle).
  * For the following cycles: regorafenib will be administered at a 80, 120 or 160 mg daily dose according to toxicity observed with the last dose used in the first cycle.
  Other Names: Stivarga
Drug: Cyclophosphamide — 50 mg per os, daily, for 6 months
  Other Names: Endoxan
Drug: Capecitabine — 625mg/m²/orally twice daily continuously for 6 months
  Other Names: Xeloda
Drug: Aspirin — 75 mg orally and daily until progression
  Other Names: Kardegic

SUMMARY:
The investigators propose a phase II clinical trial with the objective to investigate the potential clinical interest to associate regorafenib with a metronomic chemotherapy combining capecitabine, cyclophosphamide and low-dose aspirin, for the treatment of patients with metastatic colorectal cancer. The main objective of the study will be to achieve 15% of objective response rate in patients treated with multimodal metronomic chemotherapy and regorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven metastatic colorectal cancer in progression after previous standard treatments (5FU, CPT11, oxaliplatin, anti-VEGF and anti-EGFR therapy if KRAS and NRAS WT), or not considered as candidate for these treatments
* Life expectancy of at least 3 months
* Female or male with age >18 years old
* Performance status = 0 or 1 (Annex 1)
* Measurable disease defined according to RECIST v1.1 (scanner or MRI) (Annex 2)
* Adequate bone marrow, liver and renal functions.

  1. Haemoglobin ≥ 9 g/dL; absolute neutrophil count (ANC) ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L
  2. Total serum bilirubin ≤ 1.5 times upper normal value (ULN), serum alkaline phosphatase < 5 times ULN, aminotransferases (AST/ALT) ≤ 3 × ULN in absence of hepatic metastasis or ≤ 5 if presence of hepatic lesions
  3. Cockcroft glomerular filtration rate > 50 ml/min
  4. Proteinuria <2+ (dipstick urinalysis) or ≤1g/24hour
* Imaging target greater than one cm must be visible on CT,
* No contraindication to Iodine contrast media injection during CT
* For female patients of childbearing potential, negative pregnancy test within 14 days before starting the study drug. Men and women are required to use adequate birth control during the study (when applicable),
* Signed and dated informed consent,
* Ability to comply with the study protocol, in the Investigator's judgment.
* Registration in a national health care system (CMU included).

Exclusion criteria:

* Diagnosis of additional malignancy within 2 years prior to the inclusion (exception of curatively treated basal cell carcinoma of the skin and/or curatively resected in situ cervical cancer),
* Current participation in a study of an investigational agent or in the period of exclusion
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before inclusion in the trial ;
* Patient under judicial protection (curatorship, tutorship) and/or deprived of freedom,
* Planned surgical procedure within the first month of treatment or any procedure that might change the timing of regorafenib administration during the first month of treatment,
* Previous exposure to regorafenib,
* Previous exposure to other anti-angiogenic treatment than bevacizumab and aflibercept,
* Complete deficit in dihydropyrimidine deshydrogenase (DPD),
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days before start of study medication,
* Pregnant or breast-feeding subjects,
* Congestive Heart Failure ≥ New York Heart Association (NYHA) class 2, unstable angina (anginal symptomatology at rest),
* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months),
* Myocardial infarction less than 6 months before start of study drug,
* Cardiac arrhythmias requiring anti-arrhythmic therapy (beta-blockers or digoxin are permitted),
* Uncontrolled hypertension (Systolic blood pressure >150 mmHg and/or diastolic pressure >100 mmHg despite optimal medical management), or history of hypertensive crisis, or hypertensive encephalopathy
* Pleural effusion or ascites that causes respiratory compromise (≥ CTCAE grade 2 dyspnea),
* Ongoing infection >grade 2 CTCAE V5,
* Known History of human immunodeficiency virus (HIV) infection,
* Active hepatitis B or C or chronic hepatitis B or C requiring treatment with antiviral therapy,
* Subjects with seizure disorder requiring medication,
* History of organ allograft,
* Subjects with evidence or history of any bleeding diathesis, irrespective of severity,
* Any haemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study medication,
* Serious, Non-healing wound, active ulcer or untreated bone fracture,
* History of abdominal fistula, GI perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to inclusion,
* Dehydration CTCAE v5 grade ≥1,
* Known hypersensitivity to any of the study drugs, study drug classes or excipient in the formulation,
* Interstitial lung disease with ongoing signs or symptoms,
* Persistent proteinuria of CTCAE Grade 3 (>3.5 g/24 hours),
* Subject unable to swallow oral medications,
* Any malabsorption condition, unresolved toxicity higher than CTCAE (V5) Grade 1 attributed to any prior therapy/procedure excluding alopecia, hypothyroidism and oxaliplatin induced neuropathy ≤ Grade 2,
* Systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and hormonal therapy during this trial or within 3 weeks,
* Treatment with any other investigational medicinal product within 28 days prior to study entry, EXCEPT for ASPIRIN,
* Co-administration of drugs potentially interacting with regorafenib i.e. CYP3A4, CYP2C9 or UGT1A9 inducers/inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
objective response rate | From date of inclusion until end of treatment for the patient, assessed to 4 months
  The objective response rate (ORR) will be defined by RECIST v1.1 criteria as the best disease response observed during the treatment period (assessed to 4 months). ORR rate is defined as the proportion of patients whose tumor regresses or does not progress under treatment.

CONTACTS AND LOCATIONS:
Overall Officials: christophe.borg@efs.sante.fr BORG, Pr, Principal Investigator — CHU Besançon
Locations (3):
- France (3):
  - CHU de Besançon, Besançon
  - Centre georges-François Leclerc, Dijon
  - Hôpital Nord Franche-Comté, Montbéliard

IPD SHARING:
Plan to Share IPD: No